CLINICAL TRIAL: NCT02981121
Title: Hospital-based Diabetes Prevention Study in Korea: A Prospective, Multi-center, Randomized, Open-label Controlled Study
Brief Title: Hospital-based Diabetes Prevention Study in Korea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeong-taek Woo (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government); Kyungpook National University Hospital (Other); Korea University Guro Hospital (Other); Pusan National University Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Asan Medical Center (Other); Ajou University School of Medicine (Other); Severance Hospital (Other); Chonbuk National University Hospital (Other)
Responsible Party: Sponsor-Investigator, Jeong-taek Woo, Professor, Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KDPS
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: PreDiabetes
Keywords: Diabetes Prevention
MeSH Terms: conditions — Prediabetic State | interventions — Exercise; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional Management (No Intervention): A patient will receive 30 minutes of individual education from the investigator, based on the standard guidelines of the Korean Diabetes Association. And will be followed up every 6 months for 36 months.
- Life style modification (Experimental): Proceed according to the Intervention Protocol developed by the Nutrition Committee of the Korean Diabetes Association. Aim to lose more than 5% of weight within 6 months, and then aim to keep weight loss constantly. After randomization, the diabetes educator team (physician / nurse / dietician) applies the intervention program for exercise therapy and diet therapy, and manages it through online education (telephone visit) and offline education (institution visit).
  * Exercise: Moderate or abnormal exercise for more than 150 minutes per week (moderate or abnormal exercise for 30 minutes or more per day)
  * Diet remedies: Train Calorie intake, nutrient intake and Monitoring.
  Interventions: Behavioral: Exercise and Diet remedies
- Metformin (Active Comparator): After randomization, take 250 mg once a day for 2 weeks. If there is no side effect, take 500 mg once a day for 2 weeks. If there are no side effects, the maximum dose can be increased to 1000mg.
  Interventions: Drug: Metformin

INTERVENTIONS:
Behavioral: Exercise and Diet remedies
  Arms: Life style modification
Drug: Metformin
  Arms: Metformin

SUMMARY:
The investigators will study prevention effect of Life style modification on diabetes mellitus comparing with conventional management and Metformin administration.

ELIGIBILITY:
Inclusion Criteria:

1. 30<Age<71
2. BMI≥23 kg/m2
3. '75g Oral glucose tolerance 2 hours after the test Blood glucose140~199mg/dL' or 'Fasting Blood Sugar 110~125 mg/dL' or 'HbA1c 5.7%~6.4%'

Exclusion Criteria:

1. Who diagnosed with Diabetes Mellitus or Who having Drugs for Diabetes Mellitus.
2. Type 2 Diabetes Mellitus

   * Who diagnosed with Diabetes Mellitus except for maternity period.
   * Who have had drugs for Diabetes Mellitus(hypoglycemic agent or insulin) except for maternity period.
   * Fasting Glucose≥ 126 mg/dL
   * 75g Oral glucose tolerance 2 hours after the Blood glucose ≥ 200 mg/dL
   * HbA1c ≥ 6.5%
3. Who life expectancy is short.

   * Cardiac history

     * History of severe cardiovascular disease within the last 6 months (cerebral hemorrhage, stroke, myocardial infarction, angina pectoris, heart failure, etc.)
     * Systolic blood pressure >180 mmHg or Diastolic blood pressure >105 mmHg
     * aortic stenosis
     * Left bundle branch block or Third degree AV block
   * Who had been diagnosed and treated for malignant tumors including leukemia and lymphoma within the last 5 years
   * Abnormal renal function (Creatinine ≥ 1.4 mg/dL (male) or ≥ 1.3 mg/dL (female) or Urine Protein ≥ 2 +)
   * Anemia(Hematocrit <36%((male) or><33%(female)) ⑤ Cirrhosis or chronic active hepatitis (AST/ALT>３UNL)
   * Acute gastrointestinal disease (pancreatitis, infectious intestinal disease)
   * Who is scheduled major surgery within the last 3 to 6 months or just after the surgery.
   * Chronic infection (HIV, active tuberculosis, etc.)
   * Pulmonary patients who rely on oxygen or daily bronchodilators
4. Who is judged to be able to influence the clinical trial by investigator.

   * Who can not communicate
   * Those with psychiatric or cognitive impairment that may affect the compliance of the clinical trial
   * Those who do not agree to the treatment group allocation by random assignment
   * Those who participate in other studies that may interfere with the clinical trial
   * Those who lost weight by more than 10% during the past 6 months, excluding weight loss after giving birth
   * Those who can not have normal walking or exercise
   * Women who are pregnant
   * Those who are currently pregnant or who are within the last 3 months after giving birth
   * Those planning pregnancy during the clinical trial period
   * Those who have a history of drug and alcohol abuse (acute, chronic) within the last 2 years
   * Those who are not appropriate or unreliable for clinical trials at the discretion of the tester
5. Who taking medication or medical condition that may affect the diagnosis of diabetes

   * Thiazide diuretics
   * Systemic beta blockers
   * Taking Niacin for the treatment of neutropenic depression
   * Possibility of taking or injecting a systemic steroid preparation
   * Taking a serotonin reuptake inhibitor (SSRI) for weight loss purpose.
   * Taking medicine for weight loss
   * Hormone status is not appropriate during thyroid hormone replacement therapy (TSH abnormal range) (If thyroid hormone therapy is stable for more than 3 months and TSH is normal, the patient can participate in)
   * Others with other endocrine diseases (eg Cushing's syndrome, acromegaly)
   * During treatment, fasting plasma triglyceride> 600 mg / dL

Ages: 31 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Diabetes Mellitus after randomization | 36 months from the baseline
  Definition of "incidence of Diabetes Mellitus"
  * Fasting Glucose ≥126 mg/dL or
  * 75g Oral glucose tolerance test 2 hours after the Blood glucose ≥ 200 mg / dL or
  * HbA1c≥6.5%

SECONDARY OUTCOMES:
Change on HbA1c | 12, 24, 36 months from the baseline
Change on Fasting Glucose | 12, 24, 36 months from the baseline
Change on HOMA2%S | 12, 24, 36 months from the baseline
Change on HOMA2%B | 12, 24, 36 months from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kyunghee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rhee SY, Chon S, Ahn KJ, Woo JT; Korean Diabetes Prevention Study Investigators. Hospital-Based Korean Diabetes Prevention Study: A Prospective, Multi-Center, Randomized, Open-Label Controlled Study. Diabetes Metab J. 2019 Feb;43(1):49-58. doi: 10.4093/dmj.2018.0033. Epub 2018 Nov 2. PMID 30398039